CLINICAL TRIAL: NCT01017497
Title: Determination of the Optimal Planning Target Volume for Brain Metastases Treated With Stereotactic Radiosurgery
Brief Title: Optimal Planning Target Volume With Stereotactic Radiosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00017062
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-01

CONDITIONS: Brain Neoplasms; Brain Cancer
Keywords: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1mm margin (Experimental): GTV expanded by 1 mm
  Interventions: Radiation: Stereotactic Radiosurgery
- 3mm margin (Experimental): GTV expanded by 3 mm
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — PTV Diameter < 2.0 cm receives 24 Gy; PTV Diameter 2.0-3.0 cm receives 18 Gy; PTV Diameter 3.1-4.0 cm receives 15 Gy;

SUMMARY:
The purpose of this study is to estimate the rate of local control at the treated site of the metastasis as a function of 1mm versus 3mm expansion about the gross tumor volume (GTV). Each lesion, not each patient will be ranndomized to either the 1mm or 3mm margin with 40 lesions randomized to each arm.

DETAILED DESCRIPTION:
Stereotactic radiosurgery (SRS) is used either as definitive treatment alone or as a "boost" in combination with whole-brain radiotherapy (WBRT) for the treatment of brain metastases. To establish a target for SRS, the gross tumor volume (GTV) is typically defined as the contrast-enhancing volume on T1-weighted axial MRI images. In turn, the volume chosen for treatment (the planning target volume or PTV) is generated by expanding the GTV to account for microscopic extension of tumor beyond the MRI-visualized volume and deviations in patient positioning at the time of treatment., However, the optimal PTV in patients undergoing SRS of brain metastases has not been established.

This pilot randomized study of approximately 49 patients (representing a total of 80 brain lesions) should be sufficient to explore the effect of margin expansion around the GTV for brain metastases. The patients enrolled in this study will undergo radiosurgery to a planning treatment volume generated by expanding the GTV of each lesion by either a 1mm or 3mm margin. Each lesion, not each patient, will be randomized to receive either the 1mm or 3mm margin with 40 lesions randomized to each arm (a patient with multiple lesions potentially could have a lesion randomized to the 1mm arm and a different lesion randomized to the 3mm arm). The primary outcome of 12-month local recurrence and the secondary outcome of the rate of radionecrosis at the SRS treatment site will be lesion-specific outcomes. All other secondary outcomes will be patient-specific outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Life expectancy of at least 6 months.
* Karnofsky Performance Score greater than 70
* Graded prognostic assessment (GPA score 0.5 or greater
* 1 to 3 brain metastases unresectable
* Maximum tumor diameter no larger than 4cm

Exclusion Criteria:

* Primary lesion with radiosensitive histology (such as: small cell carcinoma, germ-cell tumors, lymphoma, leukemia, and multiple myeloma.
* Metastases in the brain stem, pons or medulla or within 5 mm of optic apparatus
* Previous cranial radiation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkpatrick, MD, PhD, Principal Investigator — Duke University Medical Center, Radiation Oncology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Optimal PTV: Optimal Planning Target Volume with Stereotactic Radiosurgery
Period: Overall Study
Arm/Group | Optimal PTV
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Optimal PTV
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 61 [26 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: 12-month Local Control Rate
Description: The 12-month local control rate is the percentage of lesions without recurrence at the lesion site 12 months after SRS. Time to local recurrence was defined as the time between SRS and local recurrence. If local recurrence did not occur, the time to local recurrence was censored at last follow-up (including deaths without local recurrence). Kaplan-Meier methods were used to describe the time to local recurrence.
Time Frame: 12 months after SRS
Population: This is a lesion-specific outcome. A patient could have 1 lesion randomized to the 1mm arm and a different lesion randomized to the 3mm arm, the total participants analyzed will not equal 49. Of the 80 lesions, 4 of 40 lesions in the 1-mm arm and 7 of 40 in the 3-mm arm had insufficient post-SRS imaging data to be included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesion
Arm/Group | 1mm Margin | 3mm Margin
Number analyzed (Participants) | 30 | 31
Number analyzed (Lesion) | 36 | 33
percentage of lesions | 91.4 [67.7 to 98.0] | 95.2 [70.7 to 99.3]

2. Secondary Outcome: Rate of Radionecrosis at SRS Treatment Site
Description: The rate of radionecrosis is defined as the proportion of lesions with an indication of radiation-associated changes but no evidence of viable tumor on follow-up imaging (and confirmed by tissue biopsy whenever possible).
Time Frame: 24 months after SRS
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of lesions
Units Other Than Participants: Lesion
Arm/Group | 1mm Margin | 3mm Margin
Number analyzed (Participants) | 30 | 31
Number analyzed (Lesion) | 36 | 33
proportion of lesions | 0.0278 [0.0007 to 0.1453] | 0.1515 [0.0511 to 0.3190]

3. Secondary Outcome: 12 Month Rate of Distant Brain Metastases
Description: The 12-month rate of distant brain metastases is defined as the percentage of participants with the appearance of new brain metastasis located away from the previously treated lesion (i.e. distant brain failure) 12 months after SRS. Time to the appearance of new brain metastasis was defined as the time between SRS and distant brain failure. Patients without new distant brain metastases as of the last follow-up were censored at the last follow-up date. Kaplan-Meier methods were used to describe the time to distant brain failure.
Time Frame: 12 month after SRS
Population: The rate of distant brain metastases is a patient-specific outcome. Of the 49 patients enrolled, six had insufficient post-SRS imaging data to be included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Optimal PTV
Number analyzed (Participants) | 43
percentage of participants | 45.7 [28.9 to 61.1]

4. Secondary Outcome: Median Overall Survival
Description: Overall survival was defined as the time in months from the start of SRS to the date of death or last contact if alive. Kaplan-Meier methods were used to estimate overall survival.
Time Frame: 24 months after SRS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Optimal PTV
Number analyzed (Participants) | 49
months | 10.6 [6.1 to 14.4]

5. Secondary Outcome: Quality of Life at 3 Months After SRS as Measured by the Functional Assessment of Cancer Therapy-Brain (FACT-Br)
Description: Quality of life as measured by the change in FACT-Br scores from baseline to 3 months after SRS. The FACT-Br (version 4) is comprised of the Functional Assessment of Cancer Therapy-General (FACT-G), a 27-item core questionnaire evaluating the domains of physical, family/social, emotional and functional well-being, with the addition of 23 brain cancer specific questions. The FACT-G total score is the sum of the four FACT-G domain scores. The Brain Cancer Subscale (BrCS) is the sum of 19 brain cancer specific questions. The FACT-Br Trial Outcome Index (TOI) is the sum of the BrCS score and the physical and family/social domain scores. The FACT-Br total score is the sum of the FACT-G total score and the BrCS score. Change score = score at 3 months after SRS - score at baseline. Positive change scores indicate improved quality of life.
Time Frame: Baseline to 3 months after SRS
Population: Only 24 patients of 49 enrolled completed both the baseline and month 3 questionnaire.
Measure: Mean (Standard Error); unit: Change in score from baseline to 3 month
Arm/Group | Optimal PTV
Number analyzed (Participants) | 24
Change in score from baseline to 3 month
  FACT-G: Physical Well-being (range: 0-28) | -3.2 (1.2)
  FACT-G: Family/Social Well-being (range: 0-28) | -0.4 (0.6)
  FACT-G: Emotional Well-being (range: 0-24) | 0.6 (0.9)
  FACT-G: Functional Well-being (range: 0-28) | -1.5 (1.5)
  FACT-G: Total Score (range: 0-108) | -4.5 (3.3)
  FACT-Br: BrCS (range: 0-76) | -1.3 (3.2)
  FACT-Br: TOI (range: 0-132) | -6.0 (5.3)
  FACT-Br: Total Score (range: 0-184) | -5.8 (6.1)

6. Secondary Outcome: Cognition at 3 Months After SRS as Measured by the Mini-Mental State Exam (MMSE)
Description: Cognition as measured by the change in MMSE scores from baseline to 3 months after SRS. The MMSE is an 11-item measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall and language. The minimum score is 0 and teh maximum score is 30 with higher MMSe scores indicating better cognition. Change score = score at 3 months after SRS - score at baseline. Positive change scores indicate improved cognition.
Time Frame: Baseline to 3 months after SRS
Population: Only 24 patients of 49 enrolled completed both the baseline and month 3 questionnaire.
Measure: Mean (Standard Error); unit: Change in score from baseline to 3 month
Arm/Group | Optimal PTV
Number analyzed (Participants) | 24
Change in score from baseline to 3 month | 0.3 (0.3)

7. Secondary Outcome: Cognition at 3 Months After SRS as Measured by the Trail Making Test (TMT)
Description: Cognition as measured by the change in scores on the Trail Making Test (TMT) from baseline to 3 months after SRS. The TMT consists of two parts. Part A (TMT-A) requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for Part B (TMT-B) except the person must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). The score on each part represents the amount of time required to complete the task. Change score = score at 3 months after SRS - score at baseline. Negative change scores indicate improved cognition.
Time Frame: Baseline to 3 months after SRS
Population: Only 24 patients of 49 enrolled completed both the baseline and month 3 questionnaire.
Measure: Mean (Standard Error); unit: Change in seconds baseline to 3 months
Arm/Group | Optimal PTV
Number analyzed (Participants) | 24
Change in seconds baseline to 3 months
  TMT-A | -1.9 (3.1)
  TMT-B | -19.9 (13.7)

8. Secondary Outcome: Rate of Death Due to Neurologic Causes
Description: The rate of death due to neurologic causes is defined as the percentage of participants whose death is attributable to the progression of neurological disease.
Time Frame: 24 months after SRS
Measure: Number; unit: percentage of participants
Arm/Group | Optimal PTV
Number analyzed (Participants) | 49
percentage of participants | 0.0

ADVERSE EVENTS:
Time Frame: 24 months
Description: The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, and have been converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Arm/Group | Optimal PTV
Serious Adverse Events (participants affected / at risk) | 8/49
Other Adverse Events (participants affected / at risk) | 29/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optimal PTV (N=49)
Adrenal insufficiency (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Central nervous system necrosis (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optimal PTV (N=49)
Cushingoid (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 6
Diarrhea (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 11
Gait disturbance (General disorders) | 1
Pain (General disorders) | 1
Vulval infection (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 17
Memory impairment (Nervous system disorders) | 3
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 3
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes